CLINICAL TRIAL: NCT01743690
Title: The Use of Probiotics in Patients With Symptomatic Oral Lichen Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Mette Kirstine Keller, Assistant professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-4-2011-143
Record Dates: First submitted 2012-11-28; First posted 2012-12-06 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Oral Lichen Planus; Candida Infection
Keywords: Probiotic; Candida; Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral; Candidiasis; Torulopsis | interventions — Nystatin; fluocinolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- fluocinolone, placebo (Active Comparator): fluocinolone, placebo
  Interventions: Drug: fluocinolone
- fluocinolone, probiotic (Experimental): fluocinolone, Probiotic lactobacilli reuteri
  Interventions: Biological: Probiotic lactobacilli reuteri; Drug: fluocinolone
- Nystatin, placebo (Active Comparator): Nystatin, placebo
  Interventions: Drug: Nystatin
- nystatin, probiotic (Experimental): nystatin, Probiotic lactobacilli reuteri
  Interventions: Biological: Probiotic lactobacilli reuteri; Drug: Nystatin

INTERVENTIONS:
Biological: Probiotic lactobacilli reuteri
  Other Names: L. reuteri (DSM 17938 og ATCC PTA 5289) two times a day
  Arms: fluocinolone, probiotic; nystatin, probiotic
Drug: Nystatin
  Arms: Nystatin, placebo; nystatin, probiotic
Drug: fluocinolone
  Arms: fluocinolone, placebo; fluocinolone, probiotic

SUMMARY:
The aim is to investigate the effect of probiotic bacteria on symptoms and clinical manifestations in patients with oral lichen planus (OLP).

The hypothesis is that probiotic bacteria can favor an oral environment that reduces the risk of symptomatic candidal and bacterial infection in OLP.

The negative influence of improper oral hygiene on OLP is established and overgrowth of Candida is a common problem. Nystatin is the only topical antifungal that does not interact with other drugs and to which the majority of the candida species are susceptible. Symptomatic treatment with fluocinolone is initiated in patients without candidal infection. Probiotic bacteria can affect the microbial homeostasis by reducing the overgrowth of pathogens e.g. candida. Different probiotic species have been shown to produce antifungal substances and reduce the growth of candida albicans in vitro. The probiotic strain Lactobacillus rhamnosus has been found to reduce the salivary count of yeasts among elderly in a randomized clinical study.

The study is planned as a blinded, randomized controlled study with four parallel arms. 120 OLP patients with symptoms form the mucous membranes are included in the study and will receive nystatin or fluocinolone treatment depending on positive or negative diagnosis of candidosis. In addition, they will be assigned to either the probiotic (A) or the placebo group (B) by randomization. The groups will be encouraged to take three tablets per day (morning, noon and evening)for eight weeks. The lozenges containseither two strains of the probiotic bacterium L. reuteri (A) or placebo (B). Cytosmears, saliva sample, and saline mouth wash will be taken at baseline, after the treatment period and at follow-up visits at 8, 16, 24 weeks and 1 year. Salivary counts of the probiotic strains, the clinical manifestations and symptoms associated to OLP will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Oral Lichen Planus

Exclusion Criteria:

* Antibiotic treatment within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
recurrence of candida infections | after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mette K Keller, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark